CLINICAL TRIAL: NCT02354508
Title: A Phase IIIb Multicenter, Open-label, Single Arm Study to Evaluate the Efficacy and Safety of Pasireotide in Patients With Acromegaly Inadequately Controlled With First Generation Somatostatin Analogues
Brief Title: Pasireotide in Patients With Acromegaly Inadequately Controlled With First Generation Somatostatin Analogues
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230C2413; 2014-002630-31 (EudraCT Number)
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Acromegaly
Keywords: acromegaly; GH; IGF-1; pasireotide LAR; SOM230; first generation; somatostatin analogues; growth disorder; gigantism; Pituitary adenoma; pituitary gigantism
MeSH Terms: conditions — Acromegaly; Growth Disorders; Gigantism; Pituitary Neoplasms | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pasireotide LAR (Experimental): Patients who qualify for the core phase of the study will be treated with pasireotide LAR 40 mg initially. Patients not achieving biochemical control can be up-titrated to pasireotide LAR 60 mg.
  Interventions: Drug: Pasireotide LAR

INTERVENTIONS:
Drug: Pasireotide LAR — Pasireotide 40 mg and 60 mg. Pasireotide 20 mg which was allowed for dose decrease in case of adverse event.
  Other Names: SOM230

SUMMARY:
This is a phase IIIb multicenter, open-label; single arm study to evaluate the efficacy and safety of pasireotide LAR 40 mg and 60 mg in patients with inadequately controlled acromegaly with maximal approved doses of first generation somatostatin analogues. The study will enroll inadequately controlled patients by high doses (maximal approved) of first-generation somatostatin analogues given for at least 3 months. Patients will receive pasireotide LAR 40 mg or 60 mg during the 36 week core study phase. Patients who have completed all visits of core phase and have completed all the assessments at the core phase completion visit can move into the 32-week extension phase. Patients can continue with study treatment until pasireotide LAR is commercially available and reimbursed in their respective country or until the end of the extension phase whichever occurs first.

DETAILED DESCRIPTION:
This is a phase IIIb multicenter, open-label; single arm study to evaluate the efficacy and safety of pasireotide LAR 40 mg and 60 mg in patients with inadequately controlled acromegaly with maximal doses of first generation somatostatin analogues. The study will enroll inadequately controlled patients by high doses of first-generation somatostatin analogues given for at least 3 months.

Patients will be categorized into two groups. Group 1 consists of patients treated with octreotide LAR 30 mg from countries where octreotide LAR 40mg is approved for the treatment of acromegaly at the time of screening. These patients will start a 3-months run-in phase to receive 40mg octreotide before being considered eligible to enter the core treatment phase. After 3 months of treatment have been completed, and prior to the fourth injection a mean GH and IGF-1 will be assessed. Patients who are achieving biochemical control will be considered a screen failure and they will not qualify for the core phase of the study. They will continue treatment with octreotide LAR 40 mg outside the frame of this study.

Group 2 consists of patients treated with octreotide LAR 30 mg from countries where octreotide 40mg is NOT yet approved at the time of screening. This group also includes patients already treated with octreotide LAR 40 mg or lanreotide ATG 120 mg. Patients should have been treated with the first generation SSAs for at least 3 months prior to screening. Eligible patients can directly enter the core treatment phase of the study. A run-in phase is not required for this patient population.

In the core treatment phase patients will start treatment with pasireotide LAR 40 mg every 4 weeks. At week 12, the mean GH value and IGF-1value will be assessed. Patients who have not achieved biochemical control by week 12 and do not have any tolerability issues with pasireotide LAR 40 mg will have the dose increased to 60 mg. Patients who have achieved biochemical control by week 12 will maintain a dose of pasireotide LAR 40 mg. A mean GH value and IGF-1 value will be assessed every 12 weeks until Visit 777. At weeks 16 and 28, the investigator will be able to adjust the dose based on the achievement of biochemical control and drug tolerability. If tolerability issues occur, the dose can be decreased in 20 mg. Once the tolerability issue resolves, the patients should return to the dose previously received. Patients will be treated for a total of 36 weeks during the core phase. During this period any concomitant medication for the treatment of acromegaly is prohibited. Patients are required to complete a core phase completion visit 4 weeks after the last dose of pasireotide LAR is administered. Patients who discontinue from the core phase are also required to complete the core phase completion visit 4 weeks after receiving the last pasireotide LAR dose.

Patients who have completed all visits of core phase and have completed all the assessments at the core phase completion visit (Visit 777) can move into the extension phase. The core phase completion visit performed at Visit 777, will also be the first visit (Visit 18) of the extension phase. At Visit 18, the patients will receive the same dose of pasireotide LAR that they received at week 32 (Visit 17). At week 40 (Visit 19), the investigator will decide the treatment regimen and the pasireotide LAR dose based on the achievement of biochemical control at Visit 777. Patients achieving biochemical control at the end of the core phase will continue pasireotide LAR monotherapy at the same dose of the core phase. Patients who are uncontrolled at the end of the core phase will continue pasireotide LAR 60 mg and they will be allowed to receive concomitant treatment with medications used to treat acromegaly based on the investigator's clinical judgment. GH and IGF-1 levels will be assessed every 12 weeks until week 72. At weeks 52 and 64, the investigator will be able to adjust the dose of pasireotide LAR and the regimen of the concomitant medication used to acromegaly based on the patients achievement of biochemical control and drug tolerability. Patients will be treated for a total of 32 weeks in the extension phase and receive the last dose of study treatment at week 68 (Visit 26). Patients are required to complete an extension phase completion visit (Visit 778) 4 weeks after the last dose of pasireotide LAR is administered. Patients who prematurely discontinue from the extension phase are also required to complete the extension phase completion visit (Visit 778) 4 weeks after receiving the last dose of pasireotide LAR.

After discontinuation from the study or completion of study treatment either at the core phase or extension phase of the study, all patients will be followed for safety for 12 weeks (84 days) after the last study drug administration. This visit can be performed by phone, a study visit for follow-up is not mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients ≥18 years
* Patients with confirmed diagnosis of inadequately controlled acromegaly (mean GH concentration ≥1 μg/L and sex- and age-adjusted IGF-1 >1.3 x ULN)
* Patients treated with octreotide LAR (30 mg or 40 mg) or lanreotide ATG (120 mg) monotherapy for at least 3 months prior to screening

Exclusion Criteria:

* Concomitant treatment with other medications reducing GH and or IGF-1, unless discontinued 3 months prior to screening
* Patients with compression of the optic chiasm requiring surgical intervention
* Diabetic patients with HbA1c >8% at screening
* Patients who are hypothyroid and not on adequate replacement therapy
* Patients with symptomatic cholelithiasis and acute or chronic pancreatitis
* Patients with clinically significant valvular disease
* Patients with risk factors for torsade de pointes (TdP)
* Hypokalaemia, hypomagnesaemia, uncontrolled hypothyroidism, family history of long QT syndrome or concomitant medications with known risk of TdP
* Patients with congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, history of acute MI less than one year prior to study entry or clinically significant impairment in cardiovascular function.
* Concomitant disease(s) that could prolong the QT interval such as autonomic neuropathy (caused by diabetes or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Patients with liver disease or ALT/AST > 2.0 X ULN, serum bilirubin >2.0 X ULN - Presence of Hepatitis B surface antigen or Hepatitis C antibody test
* Patients with serum creatinine >2.0 X ULN
* Patients with WBC <3 X 109/L; Hb 90% < LLN; PLT <100 X 109/L
* Patients with active or suspected acute or chronic uncontrolled infection
* Patients who have undergone major surgery/surgical therapy within 4 weeks prior to screening
* Patients with active malignant disease within the last five years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)
* Patients with abnormal coagulation (PT and/or APTT elevated by 30% above normal limits) or patients receiving anticoagulants that affect PT (prothrombin time) or APTT (activated partial thromboplastin time)
* History of syncope or family history of idiopathic sudden death
* History of immunocompromise, including a positive HIV test result (ELISA and Western blot)
* Known hypersensitivity to somatostatin analogues or any other component of pasireotide LAR
* Patients who have a history of alcohol or drug abuse in the 6 month period prior to receiving pasireotide
* Patients who have given a blood donation (of 400 ml or more) within 2 months before receiving pasireotide
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Patients with any current or prior medical condition interfering with the conduct of the study or the evaluation of the study results
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study.
* Sexually active males unless they use a condom during intercourse while taking drug and for 3 months following last dose of pasireotide
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and 3 months following the last dose of pasireotide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (47):
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro, Brazil
- Novartis Investigative Site, Sofia, Bulgaria
- China (3):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Chengdu, Sichuan
- Colombia (2):
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Bogotá
- France (8):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Hungary (2):
  - Novartis Investigative Site, Szeged, HUN
  - Novartis Investigative Site, Budapest
- Italy (8):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Malaysia (2):
  - Novartis Investigative Site, Pulau Pinang
  - Novartis Investigative Site, Wilayah Persekutuan
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Durango
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (2):
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gadelha M, Bex M, Colao A, Pedroza Garcia EM, Poiana C, Jimenez-Sanchez M, Yener S, Mukherjee R, Bartalotta A, Maamari R, Raverot G. Evaluation of the Efficacy and Safety of Switching to Pasireotide in Patients With Acromegaly Inadequately Controlled With First-Generation Somatostatin Analogs. Front Endocrinol (Lausanne). 2020 Feb 3;10:931. doi: 10.3389/fendo.2019.00931. eCollection 2019. PMID 32117045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned 112 participants and analyzed 123 participants. For Participant Flow/Baseline Characteristics Tables, Total = Participants in the Pasireotide LAR arm.
Pre-assignment Details: Participants were allocated to Group 1 or Group 2 based on previously received first generation Somatostatin analog (SSA).
Groups:
- Lanreotide 120 mg: Participants were treated with lanreotide 120mg and assigned to Group 2 (before starting on Pasireotide in the Core phase).
- Octreotide 30 mg: Participants were treated with octreotide 30 mg and assigned to Group 2 (before starting on Pasireotide in the Core phase). .
- Octreotide 40 mg: Participants were treated with octreotide 40 mg and assigned to either Group 1 (if 40mg octreotide was approved in the country) or Group 2 if 40mg octreotide was not approved in the country (before starting on Pasireotide in the Core phase).
Period: Period 1: Core Phase
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg
Started | 41 | 29 | 53
Completed (Completed 36 week (wk) Core phase) | 39 | 27 | 47
Not Completed | 2 | 2 | 6
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2
Period: Period 2: Extension Phase
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg
Started | 26 (not all patients who completed the Core phase went into the Extension phase) | 23 (not all patients who completed the Core phase went into the Extension phase) | 39 (not all patients who completed the Core phase went into the Extension phase)
Completed (Completed 72 week extension phase) | 20 | 19 | 36
Not Completed | 6 | 4 | 3
Not completed — Unsatisfactory therapeutic effect | 1 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 5 | 0 | 1
Period: Period 3: Post-treatment Follow up Phase
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg
Started (Entered post-treatment follow up) | 26 | 23 | 39
Entered Post-treatment f/up Discontinued | 4 (Entered post-treatment follow-up, discontinued) | 3 (Entered post-treatment follow-up, discontinued) | 3 (Entered post-treatment follow-up, discontinued)
Completed (Entered post-treatment follow-up, completed) | 22 (Entered post-treatment follow-up, completed) | 20 (Entered post-treatment follow-up, completed) | 36 (Entered post-treatment follow-up, completed)
Not Completed | 4 | 3 | 3
Not completed — Unsatisfactory therapeutic effect | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): comprised all patients who had signed informed consent and had been treated with at least one dose of study medication (pasireotide LAR) after enrollment into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg | Total
Number analyzed (Participants) | 41 | 29 | 53 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.02) | 41.6 (12.89) | 46.6 (11.63) | 43.8 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 25 | 62
  Male | 22 | 11 | 28 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 34 | 14 | 30 | 78
  Black | 0 | 1 | 0 | 1
  Asian | 1 | 7 | 3 | 11
  Native American | 2 | 0 | 1 | 3
  Other | 4 | 7 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36 by Previous Treatment and Overall
Description: Percentage of participants who achieved biochemical control defined as GH <1μg/L and IGF-1 <ULN at week 36.
Time Frame: Week 36
Population: Full Analysis Set (FAS) comprised all patients who had signed informed consent and had been treated with at least one dose of study medication (pasireotide LAR) after enrollment into the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR Overall: This is the sum total of participants in under the previous treatments: lanreotide 120 mg, octreotide 30 mg or octreotide 40 mg.
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg | Pasireotide LAR Overall
Number analyzed (Participants) | 41 | 29 | 53 | 123
Percentage of participants | 14.6 [5.57 to 29.17] | 13.8 [3.89 to 31.66] | 15.1 [6.75 to 27.59] | 14.6 [8.91 to 22.14]

2. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36 for Participants Up-titrated to Pasireotide LAR 60 mg
Description: Percentage of participants who achieved biochemical control defined as GH <1μg/L and IGF-1 <ULN at week 36, for participants who had been up-titrated with pasireotide LAR 60 mg.
Time Frame: Week 36
Population: Full Analysis Set (FAS) comprised all patients who had signed informed consent and had been treated with at least one dose of study medication (pasireotide LAR) after enrollment into the study. For these patients the Pasireotide LAR dose was uptitrated to 60 mg before Week 36.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Up-titrated to Pasireotide LAR 60 mg: This is the subset of participants in the FAS who started treatment with 40 mg pasireotide LAR in the core phase and were up-titrated to pasireotide LAR 60 mg.
Arm/Group | Up-titrated to Pasireotide LAR 60 mg
Number analyzed (Participants) | 90
Percentage of participants | 6.7 [2.49 to 13.95]

3. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36
Description: Percentage of participants who achieved biochemical control defined as GH <1μg/L and IGF-1 <ULN at week 36.
Time Frame: Wek 36
Population: Per-Protocol Set (PPS): consisted of a subset of the patients in the FAS who were compliant with requirements of the clinical study protocol. The protocol deviations criteria were defined prior to database lock. Per-protocol analysis was performed during the core phase, but not during the extension phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 102
Percentage of participants | 15.7 [9.24 to 24.22]

4. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36
Description: Percentage of patients who achieved biochemical control defined as GH <1μg/L and IGF-1 <ULN at week 36, by previous treatment, type of therapy and overall.
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR Monotherapy: Participants received pasireotide LAR only
- Pasireotide With Concomitant Medication: Participants received pasireotide along with other concomitant medications.or octreotide 40 mg.
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg | Pasireotide LAR Monotherapy | Pasireotide With Concomitant Medication | Pasireotide LAR Overall
Number analyzed (Participants) | 26 | 23 | 39 | 76 | 12 | 88
Percentage of participants | 7.7 [0.95 to 25.13] | 13.0 [2.78 to 33.59] | 20.5 [9.30 to 36.46] | 17.1 [9.43 to 27.47] | 0.0 [0.00 to 26.46] | 14.8 [8.11 to 23.94]

5. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36 for Participants Up-titrated to Pasireotide LAR 60 mg
Description: as for outcome 2
Time Frame: Week 36
Population: Full Analysis Set (FAS) comprised all patients who had signed informed consent and had been treated with at least one dose of study medication (pasireotide LAR) after enrollment into the study. For these patients the Pasireotide LAR dose was uptitrated to 60 mg any time during the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Up-titrated to Pasireotide LAR 60 mg: This is the subset of participants in the Extension FAS who started treatment with 40 mg pasireotide LAR in the extension phase and were up-titrated to pasireotide LAR 60 mg.
Arm/Group | Up-titrated to Pasireotide LAR 60 mg
Number analyzed (Participants) | 70
Percentage of participants | 5.9 [1.63 to 14.38]

6. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36 Overall by Baseline Diabetic Status
Description: Percentage of participants who achieved biochemical control defined as GH <1μg/L and IGF-1 <ULN at week 36, overall by baseline diabetic status.
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 88
Percentage of participants
  Diabetic: number analyzed (Participants) | 43
  Diabetic | 14.0 [5.30 to 27.93]
  Pre-diabetic: number analyzed (Participants) | 36
  Pre-diabetic | 19.4 [8.19 to 36.02]
  Non-diabetic: number analyzed (Participants) | 9
  Non-diabetic | 0.0 [0.00 to 33.63]

7. Primary Outcome: Core Phase: Percentage of Participants With Mean GH < 1 g/L and IGF-1 < ULN at Week 36 by Previous Treatment and Overall - LOCF
Description: Percentage of participants who achieved biochemical control defined as GH <1μg/L and IGF-1 <ULN at week 36, by previous treatment and overall - last observation carried forward (LOCF)
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg | Pasireotide LAR Overall
Number analyzed (Participants) | 41 | 29 | 53 | 123
Percentage of participants | 14.6 [5.57 to 29.17] | 13.8 [3.89 to 31.66] | 17.0 [8.07 to 29.80] | 15.4 [9.56 to 23.07]

8. Secondary Outcome: Core Phase: Change in Mean Growth Hormone (GH) Values From Baseline to Week 36
Description: Core phase - Changes in mean GH from study baseline to week 36.
Time Frame: Baseline, week 36
Population: FAS comprised all patients who had signed informed consent and had been treated with at least one dose of study medication (pasireotide LAR) after enrollment into the study.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg | Pasireotide LAR Overall
Number analyzed (Participants) | 41 | 29 | 53 | 123
percentage change | -7.7 (19.51) | -8.5 (24.41) | -2.9 (4.21) | -6.0 (17.10)

9. Secondary Outcome: Core Phase: Change in Standardized IGF-1 Values From Baseline to Week 36
Description: Core phase - Changes in standardized IGF-1 from study baseline to week 36.
Time Frame: Baseline, week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lanreotide 120 mg | Octreotide 30 mg | Octreotide 40 mg | Pasireotide LAR Overall
Number analyzed (Participants) | 41 | 29 | 53 | 123
percentage change | -1.1 (1.18) | -0.8 (0.78) | -1.1 (1.39) | -1.0 (1.18)

10. Secondary Outcome: Core Phase: Percentage of Participants With Mean GH <1 μg/L and IGF-1 <ULN
Description: Percentage of participants achieving GH <1 μg/L and IGF-1 <ULN at weeks 12 and 24 overall and by GH level at screening.
Time Frame: Week 12, Week 24, Week 36
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR (run-in Phase): Participants who were part of the run-in phase, i.e. group 1)
Arm/Group | Pasireotide LAR (run-in Phase) | Pasireotide LAR Overall
Number analyzed (Participants) | 17 | 123
Percentage of participants
  Week 12: GH: ≥ 1 - ≤ 2.5 μg/L @ screening: number analyzed (Participants) | 4 | 28
  Week 12: GH: ≥ 1 - ≤ 2.5 μg/L @ screening | 25.0 [0.63 to 80.59] | 28.6 [13.22 to 48.67]
  Week 24: GH: ≥ 1 - ≤ 2.5 μg/L @ screening: number analyzed (Participants) | 4 | 28
  Week 24: GH: ≥ 1 - ≤ 2.5 μg/L @ screening | 25.0 [0.63 to 80.59] | 39.3 [21.50 to 59.42]
  Week 36: GH: ≥ 1 - ≤ 2.5 μg/L @ screening: number analyzed (Participants) | 4 | 28
  Week 36: GH: ≥ 1 - ≤ 2.5 μg/L @ screening | 25.0 [0.63 to 80.59] | 42.9 [24.46 to 62.82]
  Week 12: GH: > 2.5 μg/L @ screening: number analyzed (Participants) | 13 | 94
  Week 12: GH: > 2.5 μg/L @ screening | 7.7 [0.19 to 36.03] | 5.3 [1.75 to 11.98]
  Week 24: GH: > 2.5 μg/L @ screening: number analyzed (Participants) | 13 | 94
  Week 24: GH: > 2.5 μg/L @ screening | 7.7 [0.19 to 36.03] | 5.3 [1.75 to 11.98]
  Week 36: GH: > 2.5 μg/L @ screening: number analyzed (Participants) | 13 | 94
  Week 36: GH: > 2.5 μg/L @ screening | 7.7 [0.19 to 36.03] | 6.4 [2.38 to 13.38]
  Week 12: GH: Missing: number analyzed (Participants) | 0 | 1
  Week 12: GH: Missing |  | 0.0 [0.00 to 97.50]
  Week 24: GH: Missing: number analyzed (Participants) | 0 | 1
  Week 24: GH: Missing |  | 0.0 [0.00 to 97.50]
  Week 36: GH: Missing: number analyzed (Participants) | 0 | 1
  Week 36: GH: Missing |  | 0.0 [0.00 to 97.50]

11. Secondary Outcome: Core Phase: Percentage of Participants With IGF-1 <ULN Overall by GH Level at Screening
Description: Percentage of participants achieving IGF-1 <ULN at weeks 12, 24 & 36.
Time Frame: Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- GH: ≥1 - ≤ 2.5 μg/L; GH: > 2.5 μg/L: These Participants had this GH level at screening
- GH: Missing: These Participants were missing GH levels at screening
- Pasireotide LAR Overall: This is the total sum of participants with at screening with various or missing GH levels
Arm/Group | GH: ≥1 - ≤ 2.5 μg/L | GH: > 2.5 μg/L | GH: Missing | Pasireotide LAR Overall
Number analyzed (Participants) | 28 | 94 | 1 | 123
Percentage of participants
  Week 12 | 35.7 [18.64 to 55.93] | 16.0 [9.22 to 24.95] | 0.0 [0.00 to 97.50] | 20.3 [13.61 to 28.52]
  Week 24 | 42.9 [24.46 to 62.82] | 23.4 [15.29 to 33.26] | 0.0 [0.00 to 97.50] | 27.6 [19.96 to 36.43]
  Week 36 | 50.0 [30.65 to 69.35] | 25.5 [17.09 to 35.57] | 0.0 [0.00 to 97.50] | 30.9 [22.88 to 39.86]

12. Secondary Outcome: Core Phase: Percentage of Participants With Mean GH <1 μg/L and IGF-1 <ULN Overall by Baseline Diabetic Status
Description: Core phase - Percentage of patients achieving GH <1μg/L at week 12, 24, 36 overall and by GH level at screening.
Time Frame: Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Diabetic: Participants who were diabetic in the Pasireotide LAR overall group
- Pre-diabetic: Participants who were pre-diabetic in the Pasireotide LAR overall group
- Non-diabetic: Participants who were non-diabetic in the Pasireotide LAR overall group
Arm/Group | Diabetic | Pre-diabetic | Non-diabetic
Number analyzed (Participants) | 52 | 60 | 11
Percentage of participants
  Week 12 | 13.5 [5.59 to 25.79] | 10.0 [3.76 to 20.51] | 0.0 [0.00 to 28.49]
  Week 24 | 13.5 [5.59 to 25.79] | 13.3 [5.94 to 24.59] | 9.1 [0.23 to 41.28]
  Week 36 | 15.4 [6.88 to 28.08] | 16.7 [8.29 to 28.52] | 0.0 [0.00 to 28.49]

13. Secondary Outcome: Core Phase: Change From Baseline in Scores as Measured by Acromegaly Quality of Life (AcroQoL)
Description: Evaluation of effect of pasireotide LAR on Health Related Quality of Life (HRQoL) was assessed using AcroQoL, an acromegaly-specific quality of life instrument. The AcroQol instrument is comprised of 22 questions divided into two scales: one evaluating physical aspects (8 items) and the other that addresses psychological aspects (14 items). The psychological scale can also be further divided into subscale that evaluates physical appearance and the other subscale focused on the impact of the disease on personal relationships of the patient (7 items each). Each of the questions has a 5-item Likert scale. For each dimension the scores range from 0-4 with 0 being the lowest impact and 4 being the most severe.
Time Frame: Baseline, Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pasireotide LAR Overall - AcroQOL Total Scores; Pasireotide LAR Overall - AcroQOL Physical Sub-scores; Pasireotide LAR Overall - AcroQOL Psychological Sub-scores; Pasireotide LAR Overall - AcroQOL Psycho/Appearance Sub-scores; Pasireotide LAR Overall-AcroQOL Psycho/Pers Relatns Sub-scores: This is the sum total of participants in under the previous treatments: lanreotide 120 mg, octreotide 30 mg or octreotide 40 mg.
Arm/Group | Pasireotide LAR Overall - AcroQOL Total Scores | Pasireotide LAR Overall - AcroQOL Physical Sub-scores | Pasireotide LAR Overall - AcroQOL Psychological Sub-scores | Pasireotide LAR Overall - AcroQOL Psycho/Appearance Sub-scores | Pasireotide LAR Overall-AcroQOL Psycho/Pers Relatns Sub-scores
Number analyzed (Participants) | 123 | 123 | 123 | 123 | 123
scores on a scale
  Week 12: number analyzed (Participants) | 120 | 120 | 120 | 120 | 118
  Week 12 | 4.5 (9.52) | 5.3 (12.93) | 4.1 (10.05) | 6.5 (12.43) | 1.9 (12.04)
  Week 24: number analyzed (Participants) | 118 | 118 | 118 | 118 | 117
  Week 24 | 4.7 (9.88) | 5.8 (12.26) | 4.0 (10.72) | 7.2 (14.44) | 0.9 (10.70)
  Week 36: number analyzed (Participants) | 110 | 110 | 109 | 110 | 108
  Week 36 | 4.6 (10.14) | 5.4 (13.00) | 4.3 (11.02) | 7.0 (15.33) | 1.8 (10.69)

14. Secondary Outcome: Core Phase: Percentage of Participants Reporting Levels 0 - 4 by Dimensions of Acromegaly Symptoms
Description: Symptoms of acromegaly were collected at various visits. The measurement was to be provided on a scale of 1-15 including half sizes. Investigators asked the participants to score the following symptoms of acromegaly: headache, fatigue, perspiration, paresthesias, osteoarthralgia according to a five-point score scale (0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe).
Time Frame: Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Groups:
- Pasireotide LAR Overall - Acromegaly Symptom: Headache; Pasireotide LAR Overall - Acromegaly Symptom: Fatigue; Pasireotide LAR Overall - Acromegaly Symptom: Perspiration; Pasireotide LAR Overall - Acromegaly Symptom: Osteoarthralgia; Pasireotide LAR Overall - Acromegaly Symptom: Paresthesiae: This is the sum total of participants in under the previous treatments: lanreotide 120 mg, octreotide 30 mg or octreotide 40 mg.
Arm/Group | Pasireotide LAR Overall - Acromegaly Symptom: Headache | Pasireotide LAR Overall - Acromegaly Symptom: Fatigue | Pasireotide LAR Overall - Acromegaly Symptom: Perspiration | Pasireotide LAR Overall - Acromegaly Symptom: Osteoarthralgia | Pasireotide LAR Overall - Acromegaly Symptom: Paresthesiae
Number analyzed (Participants) | 123 | 123 | 123 | 123 | 123
Percentage of participants
  Week 12: Non/absent: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 12: Non/absent | 56.9 | 37.4 | 56.9 | 43.1 | 69.1
  Week 12: Mild: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 12: Mild | 24.4 | 26.8 | 26.8 | 27.6 | 15.4
  Week 12: Moderate: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 12: Moderate | 14.6 | 18.7 | 8.1 | 14.6 | 5.7
  Week 12: Severe: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 12: Severe | 0.8 | 8.9 | 3.3 | 8.9 | 4.9
  Week 12: Very severe: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 12: Very severe | 0.0 | 4.9 | 1.6 | 2.4 | 1.6
  Week 12: Not done: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 12: Not done | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 24: Non/absent: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 24: Non/absent | 59.3 | 46.3 | 64.2 | 47.2 | 72.4
  Week 24: Mild: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 24: Mild | 27.6 | 20.3 | 21.1 | 26.8 | 13.8
  Week 24: Moderate: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 24: Moderate | 8.1 | 17.9 | 8.9 | 14.6 | 7.3
  Week 24: Severe: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 24: Severe | 1.6 | 7.3 | 1.6 | 3.3 | 0.8
  Week 24: Very severe: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 24: Very severe | 0.0 | 4.9 | 0.8 | 4.9 | 2.4
  Week 24: Not done: number analyzed (Participants) | 119 | 119 | 119 | 119 | 119
  Week 24: Not done | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 36: Non/absent: number analyzed (Participants) | 113 | 113 | 113 | 113 | 113
  Week 36: Non/absent | 63.4 | 47.2 | 61.8 | 47.2 | 69.1
  Week 36: Mild: number analyzed (Participants) | 113 | 113 | 113 | 113 | 113
  Week 36: Mild | 17.1 | 23.6 | 18.7 | 26.8 | 14.6
  Week 36: Moderate: number analyzed (Participants) | 113 | 113 | 113 | 113 | 113
  Week 36: Moderate | 9.8 | 13.0 | 7.3 | 12.2 | 5.7
  Week 36: Severe: number analyzed (Participants) | 113 | 113 | 113 | 113 | 113
  Week 36: Severe | 1.6 | 4.9 | 4.1 | 3.3 | 1.6
  Week 36: Very severe: number analyzed (Participants) | 113 | 113 | 113 | 113 | 113
  Week 36: Very severe | 0.0 | 3.3 | 0.0 | 2.4 | 0.8
  Week 36: Not done: number analyzed (Participants) | 113 | 113 | 113 | 113 | 113
  Week 36: Not done | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

15. Secondary Outcome: Core Phase: Percentage of Participants With Acromegaly Shift Symptoms From Baseline to Most Extreme Post-baseline
Description: as for outcome 14
Time Frame: Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Groups:
- Pasireotide LAR Overall - Acromegaly Symptom: Paresthsiae: This is the sum total of participants in under the previous treatments: lanreotide 120 mg, octreotide 30 mg or octreotide 40 mg
Arm/Group | Pasireotide LAR Overall - Acromegaly Symptom: Headache | Pasireotide LAR Overall - Acromegaly Symptom: Fatigue | Pasireotide LAR Overall - Acromegaly Symptom: Perspiration | Pasireotide LAR Overall - Acromegaly Symptom: Osteoarthralgia | Pasireotide LAR Overall - Acromegaly Symptom: Paresthsiae
Number analyzed (Participants) | 123 | 123 | 123 | 123 | 123
Percentage of participants
  Baseline (BL): Non/absent: number analyzed (Participants) | 51 | 45 | 53 | 41 | 67
  Baseline (BL): Non/absent | 41.5 | 36.6 | 43.1 | 33.3 | 54.5
  BL: Mild: number analyzed (Participants) | 31 | 23 | 31 | 26 | 31
  BL: Mild | 25.2 | 17.8 | 25.2 | 21.1 | 25.2
  BL: Moderate: number analyzed (Participants) | 23 | 32 | 23 | 32 | 13
  BL: Moderate | 18.7 | 26.0 | 18.7 | 26.0 | 10.6
  BL: Severe: number analyzed (Participants) | 11 | 17 | 11 | 20 | 11
  BL: Severe | 7 | 13.8 | 8.9 | 16.3 | 8.9
  BL: Very severe: number analyzed (Participants) | 7 | 6 | 5 | 4 | 1
  BL: Very severe | 5.7 | 4.9 | 4.1 | 3.3 | 0.8
  BL: Not done: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  BL: Total | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Most extr post-BL:tot Non/absent: number analyzed (Participants) | 45 | 32 | 46 | 33 | 58
  Most extr post-BL:tot Non/absent | 36.6 | 26.0 | 37.4 | 26.8 | 47.2
  Most extr. post-BL: total Mild: number analyzed (Participants) | 38 | 28 | 36 | 32 | 34
  Most extr. post-BL: total Mild | 30.9 | 22.8 | 29.3 | 26.0 | 27.6
  Most extr. post-BL: total Mod.: number analyzed (Participants) | 25 | 28 | 25 | 30 | 16
  Most extr. post-BL: total Mod. | 20.3 | 22.8 | 20.3 | 24.4 | 13.0
  Most extr. post-BL: total Severe: number analyzed (Participants) | 12 | 19 | 9 | 18 | 12
  Most extr. post-BL: total Severe | 9.8 | 15.4 | 7.3 | 14.6 | 9.8
  Most extr post-BL:tot. Very severe: number analyzed (Participants) | 3 | 16 | 7 | 10 | 3
  Most extr post-BL:tot. Very severe | 2.4 | 13.0 | 5.7 | 8.1 | 2.4
  Most extr. post-BL: total Not done: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Core Phase: Change From Baseline in EQ-5D-5L Index Scores
Description: Evaluation of effect of pasireotide LAR on health status, measured by EQ-5D-5L, a valid and reliable instrument for measuring general health status. The EQ-5D-5L consists of 2 pages - the descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a 20-cm vertical, visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'. This scale is numbered from 0 to 100. 100 means the best health you can imagine.
  0 means the worst health you can imagine.
Time Frame: Baseline, Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 123
scores on a scale
  Week 12: number analyzed (Participants) | 119
  Week 12 | 0.0 (0.15)
  Week 24: number analyzed (Participants) | 118
  Week 24 | 0.0 (0.15)
  Week 36: number analyzed (Participants) | 111
  Week 36 | 0.0 (0.15)

17. Secondary Outcome: Core Phase: Change From Baseline in EQ-5D-5L VAS Assessment
Description: as for outcome 16
Time Frame: Baseline, Weeks 12, 24 & 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 123
scores on a scale
  Week 12: number analyzed (Participants) | 119
  Week 12 | 4.1 (14.91)
  Week 24: number analyzed (Participants) | 118
  Week 24 | 3.4 (13.49)
  Week 36: number analyzed (Participants) | 111
  Week 36 | 4.9 (15.24)

18. Secondary Outcome: Extension Phase: Percentage of Participants With Mean GH < 1 μg/L and IGF-1 < ULN at Weeks 48, 60 & 72 (Up-titrated to Pasireotide LAR 60 mg)
Description: Percentage of patients achieving IGF-1 <ULN at weeks 48, 60 & 72 for participants with up-titrated to Pasireotide LAR 60 mg mg
Time Frame: Weeks 48, 60 & 72
Population: Extension Full Analysis Set (Extension FAS) included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Up-titrated to Pasireotide LAR 60 mg
Number analyzed (Participants) | 70
Percentage of participants
  Week 48 | 5.8 [1.60 to 14.18]
  Week 60 | 7.1 [2.36 to 15.89]
  Week 72 | 5.7 [1.58 to 13.99]

19. Secondary Outcome: Extension Phase: Percentage of Participants With Mean GH < 1 μg/L and IGF-1 < ULN at Weeks 48, 60 and 72 (Overall by Baseline Diabetic Status)
Description: Percentage of participants achieving IGF-1 <ULN at week 46, 60 and 72 overall by baseline diabetic status
Time Frame: Weeks 48, 60, 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR Overall: These are the participants in the extension phase who received Pasireotide LAR
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 88
Percentage of participants
  Week 48: Diabetic: number analyzed (Participants) | 43
  Week 48: Diabetic | 11.6 [3.89 to 25.08]
  Week 60: Diabetic: number analyzed (Participants) | 43
  Week 60: Diabetic | 11.6 [3.89 to 25.08]
  Week 72: Diabetic: number analyzed (Participants) | 43
  Week 72: Diabetic | 11.6 [3.89 to 25.08]
  Week 48: Pre-diabetic: number analyzed (Participants) | 36
  Week 48: Pre-diabetic | 11.1 [3.11 to 26.06]
  Week 60: Pre-diabetic: number analyzed (Participants) | 36
  Week 60: Pre-diabetic | 16.7 [6.37 to 32.81]
  Week 72: Pre-diabetic: number analyzed (Participants) | 36
  Week 72: Pre-diabetic | 8.3 [1.75 to 22.47]
  Week 48: Non-diabetic: number analyzed (Participants) | 9
  Week 48: Non-diabetic | 22.2 [2.81 to 60.01]
  Week 60: Non-diabetic: number analyzed (Participants) | 9
  Week 60: Non-diabetic | 22.2 [2.81 to 60.01]
  Week 72: Non-diabetic: number analyzed (Participants) | 9
  Week 72: Non-diabetic | 22.2 [2.81 to 60.01]

20. Secondary Outcome: Extension Phase: Percentage of Participants With Mean GH < 1 μg/L at Weeks 48, 60, 72 and Overall, Pasireotide Montherapy and Pasireotide With Concomittant Medication and by GH Level at Screening
Description: Percentage of patients achieving GH <1 μg/L and IGF-1 <ULN at week 48 by treatment with pasireotide LAR alone or with concomitant medications used to treat acromegaly
Time Frame: Weeks 48, 60, 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR Monotherapy: These Participants were treated with pasireotide LAR only in the extension phase
- Pasireotide With Concomitant Mediaction: These Participants were treated with pasireotide LAR as well as other concomitant medications in the extension phase
- Pasireotide LAR Overall: This is the sum total of participants who were treated with at least one dose of pasireotide LAR in the extension phase
Arm/Group | Pasireotide LAR Monotherapy | Pasireotide With Concomitant Mediaction | Pasireotide LAR Overall
Number analyzed (Participants) | 76 | 12 | 88
Percentage of participants
  Wk48:GH: >= 1 - <= 2.5 μg/L at screen.: number analyzed (Participants) | 17 | 3 | 20
  Wk48:GH: >= 1 - <= 2.5 μg/L at screen. | 76.5 [50.10 to 93.19] | 0.0 [0.00 to 70.76] | 65.0 [40.78 to 84.61]
  Wk60:GH: >= 1 - <= 2.5 μg/L at screen.: number analyzed (Participants) | 17 | 3 | 20
  Wk60:GH: >= 1 - <= 2.5 μg/L at screen. | 70.6 [44.04 to 89.69] | 0.0 [0.00 to 70.76] | 60.0 [36.05 to 80.88]
  Wk72:GH: >= 1 - <= 2.5 μg/L at screen.: number analyzed (Participants) | 17 | 3 | 20
  Wk72:GH: >= 1 - <= 2.5 μg/L at screen. | 64.7 [38.33 to 85.79] | 0.0 [0.00 to 70.76] | 55.0 [31.53 to 76.94]
  Wk48: GH: > 2.5 μg/L at screening: number analyzed (Participants) | 59 | 9 | 68
  Wk48: GH: > 2.5 μg/L at screening | 11.9 [4.91 to 22.93] | 11.1 [0.28 to 48.25] | 11.8 [5.22 to 21.87]
  Wk60: GH: > 2.5 μg/L at screening: number analyzed (Participants) | 59 | 9 | 68
  Wk60: GH: > 2.5 μg/L at screening | 11.9 [4.91 to 22.93] | 0.0 [0.00 to 33.63] | 10.3 [4.24 to 20.07]
  Wk72: GH: > 2.5 μg/L at screening: number analyzed (Participants) | 59 | 9 | 68
  Wk72: GH: > 2.5 μg/L at screening | 11.9 [4.91 to 22.93] | 0.0 [0.00 to 33.63] | 10.3 [4.24 to 20.07]
  Week 48: Pasireotide LAR overall | 26.3 [16.87 to 37.68] | 8.3 [0.21 to 38.48] | 23.9 [15.42 to 34.14]
  Week 60: Pasireotide LAR overall | 25.0 [15.77 to 36.26] | 0.0 [0.00 to 26.46] | 21.6 [13.53 to 31.65]
  Week 72: Pasireotide LAR overall | 23.7 [14.68 to 34.82] | 0.0 [0.00 to 26.46] | 20.5 [12.60 to 30.39]

21. Secondary Outcome: Extension Phase: Change From Baseline in Scores as Measured by Acromegaly Quality of Life (AcroQoL)
Description: as for outcome 13
Time Frame: Baseline, Weeks 48, 60 & 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Pasireotide LAR Overall - AcroQOL Total Scores; Pasireotide LAR Overall - AcroQOL Physical Sub-scores; Pasireotide LAR Overall - AcroQOL Psychological Sub-scores; Pasireotide LAR Overall - AcroQOL Psycho/Appearance Sub-scores; Pasireotide LAR Overall-AcroQOL Psycho/Pers Relatns Sub-scores: This is the sum total of participants who were treated with at least one dose of pasireotide LAR in the extension phase
Arm/Group | Pasireotide LAR Overall - AcroQOL Total Scores | Pasireotide LAR Overall - AcroQOL Physical Sub-scores | Pasireotide LAR Overall - AcroQOL Psychological Sub-scores | Pasireotide LAR Overall - AcroQOL Psycho/Appearance Sub-scores | Pasireotide LAR Overall-AcroQOL Psycho/Pers Relatns Sub-scores
Number analyzed (Participants) | 88 | 88 | 88 | 88 | 88
scores on a scale
  Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Week 60: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
  Week 60 | -4.5 (0.0) | 0.0 (0.00) | -7.1 (0.00) | -3.6 (0.00) | -10.7 (0.00)
  Week 72: number analyzed (Participants) | 74 | 74 | 73 | 74 | 72
  Week 72 | 1.6 (9.72) | 0.9 (10.61) | 1.8 (10.60) | 0.8 (12.82) | 2.9 (11.82)

22. Secondary Outcome: Extension Phase: Percentage of Participants Reporting Levels 1 - 5 by Dimensions of Acromegaly Symptoms
Description: as for outcome 14
Time Frame: Weeks 48, 60 & 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Number; unit: Percentage of participants
Groups:
- Pasireotide LAR Overall - Acromegaly Symptom: Headache; Pasireotide LAR Overall - Acromegaly Symptom: Fatigue; Pasireotide LAR Overall - Acromegaly Symptom: Perspiration; Pasireotide LAR Overall - Acromegaly Symptom: Osteoarthralgia; Pasireotide LAR Overall - Acromegaly Symptom: Paresthesiae: This is the sum total of participants who were treated with at least one dose of pasireotide LAR in the extension phase
Arm/Group | Pasireotide LAR Overall - Acromegaly Symptom: Headache | Pasireotide LAR Overall - Acromegaly Symptom: Fatigue | Pasireotide LAR Overall - Acromegaly Symptom: Perspiration | Pasireotide LAR Overall - Acromegaly Symptom: Osteoarthralgia | Pasireotide LAR Overall - Acromegaly Symptom: Paresthesiae
Number analyzed (Participants) | 88 | 88 | 88 | 88 | 88
Percentage of participants
  Week 48: None/absent: number analyzed (Participants) | 81 | 81 | 81 | 81 | 81
  Week 48: None/absent | 63.6 | 59.1 | 69.3 | 53.4 | 71.6
  Week 48: Mild: number analyzed (Participants) | 81 | 81 | 81 | 81 | 81
  Week 48: Mild | 19.3 | 17.0 | 13.6 | 25.0 | 14.8
  Week 48: Moderate: number analyzed (Participants) | 81 | 81 | 81 | 81 | 81
  Week 48: Moderate | 8.0 | 12.5 | 9.1 | 9.1 | 4.5
  Week 48: Severe: number analyzed (Participants) | 81 | 81 | 81 | 81 | 81
  Week 48: Severe | 1.1 | 3.4 | 0.0 | 3.4 | 0.0
  Week 48: Very severe: number analyzed (Participants) | 81 | 81 | 81 | 81 | 81
  Week 48: Very severe | 0.0 | 0.0 | 0.0 | 1.1 | 1.1
  Week 48: Not done: number analyzed (Participants) | 81 | 81 | 81 | 81 | 81
  Week 48: Not done | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 60: None/absent: number analyzed (Participants) | 77 | 77 | 77 | 77 | 77
  Week 60: None/absent | 60.2 | 48.9 | 60.2 | 56.8 | 70.5
  Week 60: Mild: number analyzed (Participants) | 77 | 77 | 77 | 77 | 77
  Week 60: Mild | 17.0 | 20.5 | 20.5 | 14.8 | 10.2
  Week 60: Moderate: number analyzed (Participants) | 77 | 77 | 77 | 77 | 77
  Week 60: Moderate | 6.8 | 13.6 | 6.8 | 11.4 | 4.5
  Week 60: Severe: number analyzed (Participants) | 77 | 77 | 77 | 77 | 77
  Week 60: Severe | 3.4 | 4.5 | 0.0 | 3.4 | 1.1
  Week 60: Very severe: number analyzed (Participants) | 77 | 77 | 77 | 77 | 77
  Week 60: Very severe | 0.0 | 0.0 | 0.0 | 1.1 | 1.1
  Week 60: Not done: number analyzed (Participants) | 77 | 77 | 77 | 77 | 77
  Week 60: Not done | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 72: None/absent: number analyzed (Participants) | 74 | 74 | 74 | 74 | 74
  Week 72: None/absent | 56.8 | 44.3 | 61.4 | 51.1 | 67.0
  Week 72: Mild: number analyzed (Participants) | 74 | 74 | 74 | 74 | 74
  Week 72: Mild | 17.0 | 23.9 | 15.9 | 20.5 | 11.4
  Week 72: Moderate: number analyzed (Participants) | 74 | 74 | 74 | 74 | 74
  Week 72: Moderate | 8.0 | 10.2 | 6.8 | 10.2 | 5.7
  Week 72: Severe: number analyzed (Participants) | 74 | 74 | 74 | 74 | 74
  Week 72: Severe | 2.3 | 4.5 | 0.0 | 1.1 | 0.0
  Week 72: Very severe: number analyzed (Participants) | 74 | 74 | 74 | 74 | 74
  Week 72: Very severe | 0.0 | 1.1 | 0.0 | 1.1 | 0.0
  Week 72: Not done: number analyzed (Participants) | 74 | 74 | 74 | 74 | 74
  Week 72: Not done | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

23. Secondary Outcome: Extension (Ext.) Phase: Percentage of Participants With Acromegaly Shift Symptoms From Extension Baseline to Most Extreme Post-extension Baseline
Description: as for outcome 14
Time Frame: Weeks 48, 60 & 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Number; unit: Percentage of participants
Groups:
- Pasireotide LAR Overall - Acromegaly Symptom: Paresthsiae: This is the sum total of participants who were treated with at least one dose of pasireotide LAR in the extension phase
Arm/Group | Pasireotide LAR Overall - Acromegaly Symptom: Headache | Pasireotide LAR Overall - Acromegaly Symptom: Fatigue | Pasireotide LAR Overall - Acromegaly Symptom: Perspiration | Pasireotide LAR Overall - Acromegaly Symptom: Osteoarthralgia | Pasireotide LAR Overall - Acromegaly Symptom: Paresthsiae
Number analyzed (Participants) | 88 | 88 | 88 | 88 | 88
Percentage of participants
  Ext. Baseline (BL): Non/absent: number analyzed (Participants) | 61 | 50 | 60 | 46 | 70
  Ext. Baseline (BL): Non/absent | 69.3 | 56.8 | 68.2 | 52.3 | 79.5
  Ext. BL: Mild: number analyzed (Participants) | 18 | 21 | 18 | 27 | 12
  Ext. BL: Mild | 20.5 | 23.9 | 20.5 | 30.7 | 13.6
  Ext. BL: Moderate: number analyzed (Participants) | 8 | 11 | 9 | 11 | 5
  Ext. BL: Moderate | 9.1 | 12.5 | 10.2 | 12.5 | 5.7
  Ext. BL: Severe: number analyzed (Participants) | 1 | 4 | 1 | 3 | 0
  Ext. BL: Severe | 1.1 | 4.5 | 1.1 | 3.4 |
  Ext. BL: Very severe: number analyzed (Participants) | 0 | 2 | 0 | 1 | 1
  Ext. BL: Very severe |  | 2.3 |  | 1.1 | 1.1
  Ext. BL: Not done: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Ext. BL: Total | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Most extr. post-BL:tot Non/absent: number analyzed (Participants) | 41 | 45 | 48 | 38 | 59
  Most extr. post-BL:tot Non/absent | 46.6 | 51.1 | 54.5 | 43.2 | 67.0
  Most extr. post-BL: total Mild: number analyzed (Participants) | 26 | 20 | 23 | 29 | 20
  Most extr. post-BL: total Mild | 29.5 | 22.7 | 26.1 | 33.0 | 22.7
  Most extr. post-BL: total Mod.: number analyzed (Participants) | 16 | 16 | 13 | 12 | 6
  Most extr. post-BL: total Mod. | 18.2 | 18.2 | 14.8 | 13.6 | 6.8
  Most extr. post-BL: total Severe: number analyzed (Participants) | 3 | 6 | 4 | 7 | 2
  Most extr. post-BL: total Severe | 3.4 | 6.8 | 4.5 | 8.0 | 2.3
  Most extr. post-BL: tot. Very severe: number analyzed (Participants) | 2 | 1 | 0 | 2 | 1
  Most extr. post-BL: tot. Very severe | 2.3 | 1.1 |  | 2.3 | 1.1
  Most extr. post-BL: total Not done: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Extension Phase: Change From Baseline in EQ-5D-5L Index Scores
Description: as for outcome 16
Time Frame: Baseline, Weeks 48, 60 & 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 88
scores on a scale
  Week 48: number analyzed (Participants) | 0
  Week 60: number analyzed (Participants) | 1
  Week 60 | -0.1 (0.00)
  Week 72: number analyzed (Participants) | 73
  Week 72 | 0.0 (0.08)

25. Secondary Outcome: Extension Phase: Change From Baseline in EQ-5D-5L VAS Assessment
Description: as for outcome 16
Time Frame: Baseline, Weeks 48, 60 & 72
Population: Extension FAS included all the patients who received at least one dose of pasireotide LAR in the extension phase.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pasireotide LAR Overall
Number analyzed (Participants) | 88
scores on a scale
  Week 48: number analyzed (Participants) | 0
  Week 60: number analyzed (Participants) | 1
  Week 60 | -10.0 (0.0)
  Week 72: number analyzed (Participants) | 73
  Week 72 | 1.6 (9.14)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment until end of study treatment plus 84 days post treatment, up to maximum duration of 76 weeks.
Description: AE is any sign or symptom that occurs during the study treatment plus the 84 days post treatment.
  This is a single-arm study that evaluated the efficacy of Pasireotide LAR 40mmg and 60 mg. The Lanreotide and Octreotide arms were not really arms. These arms represent the drugs that the participants were on before being enrolled in the Pasireotide LAR arm.
Groups:
- Up-titrated to Pasireotide LAR 60 mg: Patients not achieving biochemical control and were up-titrated to pasireotide LAR 60 mg.
- Pasireotide LAR Overall: This is the sum total of participants in under the previous treatments in the Core phase: lanreotide 120 mg, octreotide 30 mg or octreotide 40 mg or who were treated with at least one dose of pasireotide LAR in the extension phase
Arm/Group | Up-titrated to Pasireotide LAR 60 mg | Pasireotide LAR Overall
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/123
Serious Adverse Events (participants affected / at risk) | 6/92 | 12/123
Other Adverse Events (participants affected / at risk) | 83/92 | 112/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Up-titrated to Pasireotide LAR 60 mg (N=92) | Pasireotide LAR Overall (N=123)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Up-titrated to Pasireotide LAR 60 mg (N=92) | Pasireotide LAR Overall (N=123)
Anaemia (Blood and lymphatic system disorders) | 11 | 13
Sinus bradycardia (Cardiac disorders) | 8 | 9
Abdominal distension (Gastrointestinal disorders) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 10 | 12
Diarrhoea (Gastrointestinal disorders) | 16 | 22
Nausea (Gastrointestinal disorders) | 5 | 7
Asthenia (General disorders) | 4 | 7
Fatigue (General disorders) | 4 | 8
Injection site pain (General disorders) | 2 | 4
Cholelithiasis (Hepatobiliary disorders) | 8 | 10
Hepatic steatosis (Hepatobiliary disorders) | 7 | 7
Bronchitis (Infections and infestations) | 3 | 5
Cystitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 7 | 11
Upper respiratory tract infection (Infections and infestations) | 7 | 8
Viral upper respiratory tract infection (Infections and infestations) | 7 | 11
Blood glucose increased (Investigations) | 7 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 22 | 29
Hyperglycaemia (Metabolism and nutrition disorders) | 39 | 56
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 13
Impaired fasting glucose (Metabolism and nutrition disorders) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 8
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 11 | 14
Paraesthesia (Nervous system disorders) | 6 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 11

LIMITATIONS AND CAVEATS:
The study is a single-arm study to evaluate the safety & efficacy of pasireotide LAR in patients with inadequately controlled acromegaly who were previously on somatostatin analogues: lanreotide 120 mg, octreotide 30 mg or octreotide 40 mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-08-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT02354508/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02354508/SAP_001.pdf